CLINICAL TRIAL: NCT03316456
Title: The Role of Gut Microbiota in Intestinal Barrier Damage in Acute Leukemia Patients Undergoing Inpatient Induction Chemotherapy
Brief Title: Gut Microbiota in Intestinal Barrier Damage in Acute Leukemia Patients Undergoing Inpatient Induction
Status: Completed | Type: Observational
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2017NTLS052; HM2017-21 (Other: University of Minnesota Division of Hematology, Oncology and Transplantation)
Record Dates: First submitted 2017-10-11; First posted 2017-10-20 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Chemotherapy-Induced Gut Barrier Damage; Acute Leukemia
Keywords: AL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AL Patients Undergoing Induction Chemotherapy: Adults undergoing inpatient induction chemotherapy for newly diagnosed/relapsed acute leukemia.
  Interventions: Diagnostic Test: Observational: Stool Sample Collection; Diagnostic Test: Observational: Blood Sample Collection; Diagnostic Test: Observational: Urine Sample Collection

INTERVENTIONS:
Diagnostic Test: Observational: Stool Sample Collection — Observational: Stool Sample Collection
  - Samples will be collected on the day of the first dose of chemotherapy, then subsequently every Monday, Wednesday, Friday until Day 28 of chemotherapy, death, or discharge from the hospital, whichever occurs sooner.
Diagnostic Test: Observational: Blood Sample Collection — Observational: Blood Sample Collection
  - Samples will be collected on the day of the first dose of chemotherapy, then subsequently every Monday, Wednesday, Friday until Day 28 of chemotherapy, death, or discharge from the hospital, whichever occurs sooner.
Diagnostic Test: Observational: Urine Sample Collection — Observational: Urine Sample Collection
  - Samples will be collected on the day of the first dose of chemotherapy, then subsequently every Monday, Wednesday, Friday until Day 28 of chemotherapy, death, or discharge from the hospital, whichever occurs sooner.

SUMMARY:
This is an observational study to collect stool, blood, and urine from acute leukemia patients undergoing induction chemotherapy in order to generate preliminary data regarding the association between microbiota and chemotherapy-induced gut barrier damage. This study consists of inpatient collections of blood, urine, and stool while the patients are undergoing inpatient induction therapy. Patients will not be scheduled for any additional procedures or testing beyond what is required for clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Adults (ages 18 - 99 years) undergoing inpatient induction chemotherapy for newly diagnosed or relapsed acute leukemia (myeloid or lymphoblastic).
* Any induction regimen (standard or experimental) with planned ~4 weeks of inpatient stay
* Able to provide written voluntary consent before performance of any study related procedure.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute leukemia population at the University of Minnesota
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2017-12-26 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Variation of Gut Microbiota Composition and Diversity | Three times weekly until day 28 of chemotherapy.
  Variation of gut microbiota composition and diversity, as determined by 16s rRNA sequencing of serial stool samples, during induction chemotherapy in acute leukemia patients.

SECONDARY OUTCOMES:
Variation of Gut Barrier Integrity | Three times weekly until day 28 of chemotherapy
  Variation of gut barrier integrity, as determined by serum levels of zonulin, I-FABP, and citrulline, during induction chemotherapy in acute leukemia patients

CONTACTS AND LOCATIONS:
Overall Officials: Armin Rashidi, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Rashidi A, Ebadi M, Rehman TU, Elhusseini H, Halaweish HF, Kaiser T, Holtan SG, Khoruts A, Weisdorf DJ, Staley C. Lasting shift in the gut microbiota in patients with acute myeloid leukemia. Blood Adv. 2022 Jun 14;6(11):3451-3457. doi: 10.1182/bloodadvances.2021006783. PMID 35192686
- [Derived] Rashidi A, Ebadi M, Rehman TU, Elhusseini H, Nalluri H, Kaiser T, Ramamoorthy S, Holtan SG, Khoruts A, Weisdorf DJ, Staley C. Altered microbiota-host metabolic cross talk preceding neutropenic fever in patients with acute leukemia. Blood Adv. 2021 Oct 26;5(20):3937-3950. doi: 10.1182/bloodadvances.2021004973. PMID 34478486